CLINICAL TRIAL: NCT00111020
Title: Open Label, Non-Comparative Treatment Protocol for the Use of Sorafenib in Patients With Advanced Renal Cell Carcinoma
Brief Title: Treatment Protocol for the Use of Sorafenib in Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11868
Expanded Access: Available
Record Dates: First submitted 2005-05-16; First posted 2005-05-17 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Multi kinase inhibitor: 400 mg of Sorafenib, orally, twice a day, on a continuous basis as a single agent for the treatment of advanced RCC

SUMMARY:
This treatment protocol allows doctors to treat advanced kidney cancer with an investigational drug called sorafenib, BAY43-9006, which is being studied in clinical trials for kidney cancer and other kinds of cancer. This treatment protocol is not a clinical trial in which sorafenib is compared to another equal treatment. All patients in this protocol will be treated with sorafenib. In addition, data from the patients who participate in this protocol will provide additional information about the drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced (unresectable, recurrent or metastatic) RCC
* Patients reasonably likely to benefit from treatment with sorafenib as a single agent therapy
* Patients with an ECOG performance status of 0-2
* Patients who will not require other systemic anticancer therapy (except for bisphosphonates) while taking sorafenib
* Patients with vascular diseases such as wet macular degeneration, vasculitis, or new peptic ulcer, may be enrolled but require close monitoring in accordance with established medical practice

Exclusion Criteria:

* Patients who are currently enrolled in, are eligible for, or have access to, any other sorafenib clinical trial
* Patients who have participated in any other sorafenib trial
* Patients who have had prior therapy with investigational agent(s) within the last four weeks prior to study entry
* Life expectancy of less than two months
* Patients with cardiac arrhythmias greater than grade 1 NCI CTCAE, Version 3.0
* Patients with active coronary artery disease or ischemia
* Patients with Child-Pugh class C hepatic impairment
* Patients with severe renal impairment or who require dialysis
* Patients with active uncontrolled hypertension
* Patients with recent or active bleeding diathesis

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2567 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety parameters | From signing consent to 30 days after last dose of study drug

SECONDARY OUTCOMES:
Limited radiological evaluations | At baseline, than every 8 weeks after start of sorafenib

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (265):
- United States (258):
  - Bessemer, Alabama
  - Cullman, Alabama
  - Mobile, Alabama
  - Anchorage, Alaska
  - Glendale, Arizona
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Conway, Arkansas
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Pine Bluff, Arkansas
  - Springdale, Arkansas
  - Bakersfield, California
  - Beverly, California
  - Concord, California
  - Duarte, California
  - Fountain Valley, California
  - Glendale, California
  - Highland, California
  - La Jolla, California
  - Loma Linda, California
  - Long Beach, California
  - Los Angeles, California
  - Newport Beach, California
  - Orange, California
  - Rancho Mirage, California
  - Sacramento, California
  - Salinas, California
  - San Diego, California
  - San Francisco, California
  - Stanford, California
  - Sunnyvale, California
  - Vallejo, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Glenwood Springs, Colorado
  - Lafayette, Colorado
  - Loveland, Colorado
  - Greenwich, Connecticut
  - Hartford, Connecticut
  - Middletown, Connecticut
  - New Britain, Connecticut
  - New Haven, Connecticut
  - Norwich, Connecticut
  - Southington, Connecticut
  - Stamford, Connecticut
  - Trumbull, Connecticut
  - Boca Raton, Florida
  - Daytona Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Gainesville, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Lakeland, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Ocala, Florida
  - Ocoee, Florida
  - Orlando, Florida
  - Ormond Beach, Florida
  - Panama City, Florida
  - Pensacola, Florida
  - St. Petersburg, Florida
  - Stuart, Florida
  - Tampa, Florida
  - Weston, Florida
  - Albany, Georgia
  - Atlanta, Georgia
  - Augusta, Georgia
  - Columbus, Georgia
  - Macon, Georgia
  - Tamc, Hawaii
  - Coeur d'Alene, Idaho
  - Chicago, Illinois
  - Decatur, Illinois
  - Harvey, Illinois
  - Joliet, Illinois
  - Niles, Illinois
  - Peoria, Illinois
  - Springfield, Illinois
  - Urbana, Illinois
  - Beech Grove, Indiana
  - Evansville, Indiana
  - Fishers, Indiana
  - Goshen, Indiana
  - Indianapolis, Indiana
  - Kokomo, Indiana
  - La Porte, Indiana
  - South Bend, Indiana
  - Valparaiso, Indiana
  - Ames, Iowa
  - Cedar Rapids, Iowa
  - Council Bluffs, Iowa
  - Des Moines, Iowa
  - Dubuqe, Iowa
  - Sioux City, Iowa
  - Hutchinson, Kansas
  - Lawrence, Kansas
  - Olathe, Kansas
  - Overland Park, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Baton Rouge, Louisiana
  - Houma, Louisiana
  - Lafayette, Louisiana
  - Metairie, Louisiana
  - Shreveport, Louisiana
  - Bangor, Maine
  - Scarborough, Maine
  - Annapolis, Maryland
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Chevy Chase, Maryland
  - Clinton, Maryland
  - Rockville, Maryland
  - Boston, Massachusetts
  - Jamaica Plain, Massachusetts
  - Milford, Massachusetts
  - Quincy, Massachusetts
  - Springfield, Massachusetts
  - Ann Arbor, Michigan
  - Clinton Township, Michigan
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Marquette, Michigan
  - Mount Clemens, Michigan
  - Muskegon, Michigan
  - Duluth, Minnesota
  - Minneapolis, Minnesota
  - Saint Louis Park, Minnesota
  - Willmar, Minnesota
  - Kansas City, Missouri
  - Saint Joseph, Missouri
  - Springfield, Missouri
  - St Louis, Missouri
  - Missoula, Montana
  - Lincoln, Nebraska
  - North Platte, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - Portsmouth, New Hampshire
  - Belleville, New Jersey
  - East Orange, New Jersey
  - Hackensack, New Jersey
  - Long Branch, New Jersey
  - Montclair, New Jersey
  - Morristown, New Jersey
  - New Brunswick, New Jersey
  - Newark, New Jersey
  - Phillipsburg, New Jersey
  - Summit, New Jersey
  - Albuquerque, New Mexico
  - Santa Fe, New Mexico
  - Armonk, New York
  - Bay Shore, New York
  - Buffalo, New York
  - Cooperstown, New York
  - Dunkirk, New York
  - East Syracuse, New York
  - Fresh Meadows, New York
  - Glens Falls, New York
  - Jamaica, New York
  - Johnson City, New York
  - Latham, New York
  - Mineola, New York
  - Mount Kisco, New York
  - New York, New York
  - Poughkeepsie, New York
  - Rochester, New York
  - Setauket, New York
  - Stony Brook, New York
  - The Bronx, New York
  - Utica, New York
  - Williamsville, New York
  - Burlington, North Carolina
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Hickory, North Carolina
  - Kinston, North Carolina
  - Pollocksville, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Barberton, Ohio
  - Canton, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Mayfield Heights, Ohio
  - Middletown, Ohio
  - Lawton, Oklahoma
  - Midwest City, Oklahoma
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Bend, Oregon
  - Medford, Oregon
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Bethlehem, Pennsylvania
  - Dunmore, Pennsylvania
  - East Stroudsburg, Pennsylvania
  - Harrisburg, Pennsylvania
  - Hermitage, Pennsylvania
  - Kittanning, Pennsylvania
  - Lancaster, Pennsylvania
  - Lemoyne, Pennsylvania
  - Monongahela, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pottsville, Pennsylvania
  - State College, Pennsylvania
  - Wynnewood, Pennsylvania
  - York, Pennsylvania
  - Cranston, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Florence, South Carolina
  - North Charleston, South Carolina
  - Sioux Falls, South Dakota
  - Clarksville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Arlington, Texas
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Midland, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Tyler, Texas
  - Ogden, Utah
  - Salt Lake City, Utah
  - Bennington, Vermont
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Lynchburg, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Lacey, Washington
  - Seattle, Washington
  - Tacoma, Washington
  - Vancouver, Washington
  - Yakima, Washington
  - Charleston, West Virginia
  - Huntington, West Virginia
  - Morgantown, West Virginia
  - Glendale, Wisconsin
  - Green Bay, Wisconsin
  - Madison, Wisconsin
  - Marshfield, Wisconsin
  - Milwaukee, Wisconsin
  - Wausau, Wisconsin
- Canada (7):
  - Edmonton, Alberta
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Derived] Stadler WM, Figlin RA, McDermott DF, Dutcher JP, Knox JJ, Miller WH Jr, Hainsworth JD, Henderson CA, George JR, Hajdenberg J, Kindwall-Keller TL, Ernstoff MS, Drabkin HA, Curti BD, Chu L, Ryan CW, Hotte SJ, Xia C, Cupit L, Bukowski RM; ARCCS Study Investigators. Safety and efficacy results of the advanced renal cell carcinoma sorafenib expanded access program in North America. Cancer. 2010 Mar 1;116(5):1272-80. doi: 10.1002/cncr.24864. PMID 20082451